CLINICAL TRIAL: NCT04544787
Title: A Phase 2, Partial Blind, Randomized, Placebo-controlled, Multicenter Study to Evaluate the Safety and Immunogenicity of Two Novel Live Attenuated Serotype 2 Oral Poliovirus Vaccines Candidates, in Healthy Adults Previously Vaccinated With Oral Polio Vaccine (OPV) or Inactivated Polio Vaccine (IPV), Compared With Historical Controls Given Sabin OPV2 or Placebo
Brief Title: A Phase 2 Study to Evaluate the Safety and Immunogenicity of Two Oral Poliovirus Vaccine Candidates
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pierre Van Damme (Other)
Collaborators: Bill and Melinda Gates Foundation (Other); Centers for Disease Control and Prevention (U.S. Federal Agency); PATH (Other); Celerion (Industry)
Responsible Party: Sponsor-Investigator, Pierre Van Damme, Full Professor, Universiteit Antwerpen
Organization: Universiteit Antwerpen (Other)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UAM4; 2018-001684-22 (EudraCT Number)
Record Dates: First submitted 2020-07-14; First posted 2020-09-10 (Actual); Results first posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-09

CONDITIONS: Poliomyelitis
Keywords: IPV-primed; adults; vaccination; shedding; genetic stability; safety; neurovirulence; novel polio vaccine candidates
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Intervention Model Description: In this partial-blind study participants will be randomized into one of the following groups:
  OPV-vaccinated adults:
  * 1 dose of nOPV2 candidate 1 (Group 1);
  * 2 doses of nOPV2 candidate 1 (Group 2);
  * 1 dose of nOPV2 candidate 2 (Group 3);
  * 2 doses of nOPV2 candidate 2 (Group 4);
  IPV-only vaccinated adults:
  * 2 doses of nOPV2 candidate 1 (Group 5);
  * 2 doses of nOPV2 candidate 2 (Group 6);
  * 2 doses of placebo (Group 7).
  The first 100 OPV-vaccinated participants will be randomly assigned 1:1 to Groups 3 (1 dose) and 4 (2 doses) to receive nOPV2-c2. The second 100 OPV-vaccinated participants will be randomly assigned 1:1 to Groups 1 (1 dose) and 2 (2 doses) to receive nOPV2-c1. IPV-vaccinated adults will be enrolled in parallel and randomly assigned 2:1 to Group 6 (2 doses of nOPV2-c2) or Group 7 (2 doses of placebo), until Group 6 enrollment is complete, when 2:1 randomization will be continued for Group 5 (2 doses of nOPV2-c1) and Group 7 (2 doses of placebo).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All OPV-vaccinated participants will receive one of the nOPV2 candidates candidates in a single blind manner and all IPV- vaccinated participants will receive one of the nOPV2 candidates or placebo in a double-blinded manner.
  For the study duration participants and blinded study staff responsible for safety evaluation of IPV participants will not have any information of what has been administered. As the placebo can be distinguished from the vaccine candidates in packaging and color, reception of the vaccines, dose preparation and administration will be done by a team of unblinded study personnel. Appropriate measures will be taken at the site to ensure blinding of subjects and blinded team for the duration of the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Group 1: One Dose of Novel OPV2 Candidate 1 (Experimental): Participants previously vaccinated with oral polio vaccine (OPV) received one dose of novel OPV2 candidate 1 on Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ 50% cell culture infectious dose units [CCID50]).
  Interventions: Biological: Novel OPV2 candidate 1
- Group 2: Two Doses of Novel OPV2 Candidate 1 (Experimental): Participants previously vaccinated with OPV received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 1
- Group 3: One Dose of Novel OPV2 Candidate 2 (Experimental): Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 2 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 2
- Group 4: Two Doses of Novel OPV2 Candidate 2 (Experimental): Participants previously vaccinated OPV received two doses novel OPV2 candidate 2 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 2
- Group 5: Two Doses of Novel OPV2 Candidate 1 (Experimental): Participants previously vaccinated with inactivated polio vaccine (IPV) received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 1
- Group 6: Two Doses of Novel OPV2 Candidate 2 (Experimental): Participants previously vaccinated with IPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
  Interventions: Biological: Novel OPV2 candidate 2
- Group 7: Two Doses of Placebo (Placebo Comparator): Participants previously vaccinated with IPV received two doses of placebo 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Novel OPV2 candidate 1 — Live-attenuated serotype-2 poliovirus derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells; candidate 1 (S2/cre5/S15domV/rec1/hifi3).
  Modifications included the following:
  * Changes to the viral nucleotide sequence in part of the 5'-untranslated region to improve the genetic stability of this major attenuating determinant of Sabin type-2 to avoid reversion by single nucleotide changes.
  * Two modifications in the polymerase 3D to further improve stability of the attenuation and reduce frequency of recombination events
  * Relocation of a key replication element from the 2C coding region to the 5'-untranslated region, to inhibit recombination.
  Arms: Group 1: One Dose of Novel OPV2 Candidate 1; Group 2: Two Doses of Novel OPV2 Candidate 1; Group 5: Two Doses of Novel OPV2 Candidate 1
Biological: Novel OPV2 candidate 2 — Live-attenuated serotype-2 poliovirus derived from a modified Sabin type-2 infectious cDNA clone and propagated in Vero cells; candidate 2 (S2/S15domV/CpG40).
  Modifications included the following:
  * Changes to the viral nucleotide sequence in part of the 5'-untranslated region to improve the genetic stability of this major attenuating determinant of Sabin type-2 to avoid reversion by single nucleotide changes.
  * silent non-coding modifications engineered within the capsid (VP1-4) designed to reduce replicative fitness and, potentially, to improve stability of the attenuated phenotype while also reducing transmission.
  Arms: Group 3: One Dose of Novel OPV2 Candidate 2; Group 4: Two Doses of Novel OPV2 Candidate 2; Group 6: Two Doses of Novel OPV2 Candidate 2
Biological: Placebo — sugar syrup, propylene glycol (Sirupus simplex, Propylenglycolum, European Pharmacopoeia)
  Arms: Group 7: Two Doses of Placebo

SUMMARY:
This study is designed to evaluate the safety and immunogenicity of two novel type 2 oral poliovirus vaccine (nOPV2) candidates (nOPV2 candidate 1 and nOPV2 candidate 2) in adults. The primary objectives of the study include the general safety and immunogenicity of the two candidate vaccines in healthy volunteers previously vaccinated with Sabin monovalent OPV or inactivated polio vaccine (IPV) only.

DETAILED DESCRIPTION:
Two nOPV2 vaccine candidates have been developed as attenuated serotype 2 polioviruses derived from a modified Sabin 2 infectious complementary deoxyribonucleic acid (cDNA) clone. nOPV2 Candidate 1 (S2/cre5/S15domV/rec1/hifi3) and nOPV2 Candidate 2 (S2/S15domV/CpG40) were generated by modifying the Sabin-2 ribonucleic acid (RNA) sequence to improve phenotypic stability and make the strains less prone to reversion to virulence. The novel vaccine will eventually be licensed based on 3 criteria: a similar safety profile to the currently licensed monovalent OPV2 (mOPV2) of the Sabin strain, non-inferior immunogenicity, and reduced reversion to virulence.

Due to the withdrawal of Sabin monovalent oral polio vaccine type 2 and prohibition of its use from April 2016 onward, well before the availability of nOPV2 for clinical testing, a head to head comparison of nOPV2 and mOPV2 is not possible. For these reasons, Phase 4 trials have been conducted with Sabin mOPV2 to provide control data on safety, immunogenicity, against which data for nOPV2 in subsequent Phase I and II studies will be evaluated and compared. The Phase 4 trials of Sabin mOPV2 were designed to parallel the expected design of the Phase 1 and 2 nOPV2 studies with respect to overall design, inclusion of similar study cohorts.

This study is designed to evaluate the safety and immunogenicity of two novel type 2 OPV candidates in adults before testing in young children and then infants. The study will include both OPV-vaccinated and IPV-vaccinated adults to provide safety and immunogenicity data relevant to the decision to advance to future studies with testing in children who have not been exposed to OPV2. The primary objectives of the study include the general safety and immunogenicity of the two candidate vaccines, primarily based on comparison with historical data obtained in a Phase 4 study of Sabin mOPV2 for OPV-vaccinated subjects, in order to establish non-inferior immunogenicity and acceptable safety profile. Assessment of the general safety of the 2 candidate vaccines in IPV-only vaccinated participants will be based on comparison with data from a placebo group.

The phase 4 control study (UAM1) used for the comparison in this study is registered with EudraCT (2015-003325-33). Participants were healthy adults aged 18-50 years with documented history of at least three polio vaccinations, including OPV, and were randomly assigned to either one dose or two doses of monovalent OPV2. Between January and March 2016, 100 volunteers were enrolled and randomly assigned to receive one or two doses of monovalent OPV2 (n=50 in each group).

ELIGIBILITY:
Inclusion Criteria:

1. For Groups 1, 2, 3 and 4: healthy males or females, from 18 to 50 years of age inclusive, having previously received at least 3 doses of OPV more than 12 months before the start of the study;
2. For Groups 5, 6 and 7: healthy males or females, from 18 to 50 years of age inclusive, having previously received at least 3 doses of IPV more than 12 months before the start of the study;
3. Having residence in Belgium;
4. In good physical and mental health as determined on the basis of medical history and general physical examination performed at Day 0;
5. Female subjects of childbearing potential must agree to the use of an effective method of birth control throughout the study and up to 3 months after last vaccine dose;
6. Willing to adhere to the prohibitions and restrictions specified in this protocol;
7. Informed Consent Form (ICF) and Code of Conduct signed voluntarily by the subject before any study-related procedure is performed, indicating that the subject understands the purpose of any procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. A condition that, in the opinion of the Investigator, could compromise the well-being of the subject or course of the study, or prevent the subject from meeting or performing any study requirements;
2. For Groups 5, 6 and 7: ever having received any OPV in the past;
3. Any travel to polio endemic countries or countries with evidence of recent (within last 6 months) wild or vaccine-derived poliovirus circulation during the total duration of the study;
4. Professional handling of food, catering or food production activities during the total duration of the study;
5. Having Crohn's disease or ulcerative colitis or having had major surgery of the gastrointestinal tract involving significant loss or resection of the bowel;
6. A known allergy, hypersensitivity, or intolerance to the study vaccine or the placebo, or to any of their components or to any antibiotics;
7. Any confirmed or suspected immunosuppressive or immunodeficiency condition (including human immunodeficiency virus [HIV] infection, hepatitis B or C infections or total serum immunoglobulin A [IgA] level below laboratory lower limit of normal [LLN]);
8. Will have household or professional contact with known immunosuppressed people or people without full polio vaccination (i.e. complete primary infant immunization series), e.g. babysitting during the total duration of the study;
9. Neonatal nurses or others having professional contact with children under 6 months of age during the total duration of the study;
10. Chronic administration (i.e., longer than 14 days) of immunosuppressant drugs or other immune-modifying drugs within 6 months prior to the first vaccine dose or planned use during the study. For instance, for corticosteroids, this means prednisone, or equivalent, ≥ 0.5 mg/kg/day (inhaled and topical steroids are allowed whereas intra-articular and epidural injection/administration of steroids are not allowed);
11. Presence of contraindications to administration of the study vaccine on Day 0: acute severe febrile illness deemed by the Investigator to be a contraindication for vaccination or persistent diarrhea or vomiting;
12. Indications of drug abuse or excessive use of alcohol at Day 0 (males: > 21 units/week; females > 14 units/week);
13. Being pregnant or breastfeeding. Women of childbearing potential will undergo a urine pregnancy test at each vaccination visit. Subjects with a positive pregnancy test will be excluded;
14. Participation in another clinical study within 28 days prior to entry in this study or receipt of any investigational product (drug or vaccine) other than the study vaccine within 28 days prior to the first administration of study vaccine, or planned use during the study period;
15. Administration of any vaccine other than the study vaccine within 28 days prior to the first dose of study vaccine and during the entire study period;
16. Administration of any polio vaccine within 12 months before the start of the study;
17. Having had a transfusion of any blood product or application of immunoglobulins within the 4 weeks prior to the first administration of study vaccine or during the study;
18. Subject is an employee of the Investigator or study site, with direct involvement in the proposed study or other studies under the direction of that Investigator or study site, or is a family member of an employee or the Investigator, or was a study subject in the historical control studies UAM1 or UAT1 or in the study UAM4a (NCT03430349);
19. Having a family or household member participating in the study CVIA 065 (NCT04232943) or being a study subject in the study CVIA 065.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Van Damme, Prof. MD, Principal Investigator — Centre for the evaluation of vaccination
Locations (2):
- Belgium (2):
  - Centre for the Evaluation of Vaccination, Vaccine & Infectious Disease Institute, University of Antwerp, Wilrijk, Antwerp
  - CEVAC, Center for Vaccinology, Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] De Coster I, Leroux-Roels I, Bandyopadhyay AS, Gast C, Withanage K, Steenackers K, De Smedt P, Aerssens A, Leroux-Roels G, Oberste MS, Konopka-Anstadt JL, Weldon WC, Fix A, Konz J, Wahid R, Modlin J, Clemens R, Costa Clemens SA, Bachtiar NS, Van Damme P. Safety and immunogenicity of two novel type 2 oral poliovirus vaccine candidates compared with a monovalent type 2 oral poliovirus vaccine in healthy adults: two clinical trials. Lancet. 2021 Jan 2;397(10268):39-50. doi: 10.1016/S0140-6736(20)32541-1. Epub 2020 Dec 9. PMID 33308429
- [Derived] Thompson KM, Kalkowska DA, Kidd SE, Burns CC, Badizadegan K. Trade-offs of different poliovirus vaccine options for outbreak response in the United States and other countries that only use inactivated poliovirus vaccine (IPV) in routine immunization. Vaccine. 2024 Feb 6;42(4):819-827. doi: 10.1016/j.vaccine.2023.12.081. Epub 2024 Jan 12. PMID 38218668

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 2 centers in Belgium. Two hundred and seventy-seven volunteers were screened between October 2018, and February 2019, and 250 participants were enrolled. Eligible participants were healthy adults aged 18-50 years with documented history of at least three polio vaccinations with either oral polio vaccine (OPV) or inactivated polio vaccine (IPV).
  Two novel oral polio type 2 vaccines (nOPV2) were tested: candidate 1 (nOPV2-c1) and candidate 2 (nOPV2-c2).
Pre-assignment Details: The novel OPV2-c2 candidate was prioritized so the first 100 OPV-vaccinated participants were randomly assigned 1:1 to Groups 3 and 4 to receive novel OPV2-c2. The second 100 OPV-vaccinated participants were randomly assigned 1:1 to Groups 1 and 2 to receive novel OPV2-c1. IPV-vaccinated adults were enrolled in parallel and randomly assigned 2:1 to Group 6 or Group 7 until Group 6 enrollment was complete, when 2:1 randomization was continued for Group 5 and Group 7.
Groups:
- Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received one dose of novel oral polio vaccine type 2 (nOPV2) candidate 1 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ 50% cell culture infectious dose units [CCID50]).
- Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
- Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 2 on study Day 0, administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
- Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
- Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1: Participants previously vaccinated with only IPV received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
- Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2: Participants previously vaccinated with only IPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total; approximately 10⁶ CCID50).
- Group 7: IPV-vaccinated - Two Doses of Placebo: Participants previously vaccinated with only IPV received two doses of placebo 28 days apart (Day 0 and Day 28), administered orally as six drops (0.3 mL total).
Period: Overall Study
Arm/Group | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Started | 50 | 50 | 50 | 50 | 17 | 16 | 17
Received First Dose of Vaccine | 50 | 50 | 50 | 50 | 17 | 16 | 17
Received Second Dose of Vaccine | 0 | 49 | 0 | 49 | 17 | 15 | 16
Completed (defined as completing the last study visit (Day 70)) | 50 | 50 | 50 | 50 | 17 | 16 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Groups:
- Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 1 on study Day 0.
- Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28).
- Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 2 on study Day 0.
- Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28).
- Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1: Participants previously vaccinated with only IPV received two doses of novel OPV2 candidate 1 28 days apart (Day 0 and Day 28).
- Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2: Participants previously vaccinated with only IPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28).
- Group 7: IPV-vaccinated - Two Doses of Placebo: Participants previously vaccinated with only IPV received two doses of placebo 28 days apart (Day 0 and Day 28).
- Total: Total of all reporting groups
Arm/Group | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 17 | 16 | 17 | 250
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10) | 31 (10) | 32 (10) | 34 (10) | 23 (10) | 31 (9) | 24 (9) | 29 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 29 | 28 | 32 | 11 | 13 | 14 | 149
  Male | 28 | 21 | 22 | 18 | 6 | 3 | 3 | 101
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 49 | 49 | 49 | 49 | 16 | 16 | 15 | 243
  Asian | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Other | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 5
Number of Prior OPV Vaccinations [Count of Participants; unit: Participants] — OPV-vaccinated participants could have also received IPV, but IPV participants were specifically only to have received IPV, no OPV dose.
  Participants
    None | 0 | 0 | 0 | 0 | 17 | 16 | 17 | 50
    Three | 49 | 50 | 41 | 40 | 0 | 0 | 0 | 180
    Four | 1 | 0 | 9 | 9 | 0 | 0 | 0 | 19
    Five | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Number of Prior IPV Vaccinations [Count of Participants; unit: Participants] — OPV-vaccinated participants could have also received IPV, but IPV participants were specifically only to have received IPV, no OPV dose.
  Participants
    None | 46 | 49 | 48 | 47 | 0 | 0 | 0 | 190
    One | 4 | 1 | 2 | 3 | 0 | 0 | 0 | 10
    Four | 0 | 0 | 0 | 0 | 6 | 4 | 10 | 20
    Five | 0 | 0 | 0 | 0 | 10 | 5 | 5 | 20
    Six or more | 0 | 0 | 0 | 0 | 1 | 7 | 2 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Severe Adverse Events
Description: An SAE is any untoward medical occurrence that at any dose met any of the following conditions:
  * Resulted in death;
  * Was life-threatening;
  * Required inpatient hospitalization or prolongation of existing inpatient hospitalization;
  * Resulted in persistent or significant disability/incapacity;
  * Was a congenital anomaly/birth defect;
  * Was medically important.
  A solicited AE is a pre-selected sign or symptom that occurred within 7 days after each dose, whereas unsolicited AEs were collected throughout the study. Solicited AEs included headache, fatigue, myalgia, arthralgia, paresthesia, anesthesia, paralysis, nausea, vomiting, diarrhea, abdominal pain, and fever.
  A severe AE is an AE that prevented normal everyday activities and which was not classified as an SAE.
  A related AE is an AE the investigator considered probably or possibly caused by the study vaccine, meaning that there was a reasonable temporal association or the AE was not attributable to other conditions.
Time Frame: Up to 42 days after each vaccination
Population: The total vaccinated (TV) population includes all randomized participants who received at least one dose of study vaccine.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 1 on Day 0.
Arm/Group | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 17 | 16 | 17
Participants
  Serious or Severe adverse event | 9 | 16 | 5 | 8 | 5 | 6 | 10
  Serious adverse events | 1 | 1 | 0 | 1 | 0 | 1 | 0
  Serious solicited adverse events | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serious unsolicited adverse events | 1 | 1 | 0 | 1 | 0 | 1 | 0
  Serious adverse events related to study vaccine | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Severe adverse events | 9 | 16 | 5 | 8 | 5 | 6 | 10
  Severe solicited adverse events | 1 | 2 | 1 | 2 | 1 | 1 | 2
  Severe unsolicited adverse events | 8 | 15 | 4 | 7 | 4 | 5 | 9
  Severe adverse events related to study vaccine | 1 | 2 | 1 | 2 | 2 | 5 | 4
Statistical Analysis 1: Comparison: Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 vs Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1; The number of participants with severe solicited adverse events in the OPV-vaccinated groups who received nOPV-c1 (combined Groups 1 and 2) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with severe solicited adverse events was 5 out of 100; Test type: Other; p = 0.7209, Fisher Exact
Statistical Analysis 2: Comparison: Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 vs Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2; The number of participants with severe solicited adverse events in the OPV-vaccinated groups who received nOPV-c2 (combined Groups 3 and 4) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with severe solicited adverse events was 5 out of 100; Test type: Other; p = 0.7209, Fisher Exact
Statistical Analysis 3: Comparison: Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 vs Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1; The number of participants with severe unsolicited adverse events in the OPV-vaccinated groups who received nOPV-c1 (combined Groups 1 and 2) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with severe unsolicited adverse events was 17 out of 100; Test type: Other; p = 0.3769, Fisher Exact
Statistical Analysis 4: Comparison: Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 vs Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2; The number of participants with severe unsolicited adverse events in the OPV-vaccinated groups who received nOPV-c2 (combined Groups 3 and 4) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with severe unsolicited adverse events was 17 out of 100; Test type: Other; p = 0.3083, Fisher Exact
Statistical Analysis 5: Comparison: Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 vs Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1; The number of participants with serious unsolicited adverse events in the OPV-vaccinated groups who received nOPV-c1 (combined Groups 1 and 2) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with serious unsolicited adverse events was 0 out of 100; Test type: Other; p = 0.4975, Fisher Exact
Statistical Analysis 6: Comparison: Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 vs Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2; The number of participants with serious unsolicited adverse events in the OPV-vaccinated groups who received nOPV-c2 (combined Groups 3 and 4) was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33) using the two-sided Fisher's exact test. In the UAM1 study, the number of participants with serious unsolicited adverse events was 0 out of 100; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 7: Comparison: Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 vs Group 7: IPV-vaccinated - Two Doses of Placebo; Comparison of severe solicited adverse events; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 8: Comparison: Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 vs Group 7: IPV-vaccinated - Two Doses of Placebo; Comparison of severe solicited adverse events; Test type: Other; p = 1.0000, Fisher Exact
Statistical Analysis 9: Comparison: Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 vs Group 7: IPV-vaccinated - Two Doses of Placebo; Comparison of severe unsolicited adverse events; Test type: Other; p = 0.1571, Fisher Exact
Statistical Analysis 10: Comparison: Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 vs Group 7: IPV-vaccinated - Two Doses of Placebo; Comparison of severe unsolicited adverse events; Test type: Other; p = 0.2960, Fisher Exact

2. Primary Outcome: Seroprotection Rate After a Single Dose of Novel OPV2 in Former OPV Recipients
Description: Seroprotection rate was defined as the percentage of participants with anti-type 2-specific poliovirus neutralizing antibody titers ≥ 1:8.
  Neutralizing antibodies against poliovirus type 2 were determined using the World Health Organization (WHO) standard microneutralization assay (WHO EPI GEN 93.9). The lower limit of quantitation (LLOQ) was 5.7 and the upper limit of quantitation (ULOQ) was 1448.
Time Frame: Baseline (Day 0 prior to vaccination) and Day 28
Population: Participants in the per-protocol population previously vaccinated with OPV. The per-protocol population excluded participants with missed doses or major protocol deviations considered to have a potential impact on immunogenicity from the time of the deviation and at all time points thereafter.
  This endpoint was analyzed after one dose of nOPV hence Groups 1 and 2 and Groups 3 and 4 are combined for analysis, as specified in the study protocol.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 1 on study Day 0.
- Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received one dose of novel OPV2 candidate 2 on study Day 0.
Arm/Group | Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 | Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2
Number analyzed (Participants) | 98 | 98
percentage of participants
  Day 0 (pre-vaccination) | 99 [94 to 100] | 94 [87 to 98]
  Day 28: number analyzed (Participants) | 96 | 98
  Day 28 | 100 [96 to 100] | 100 [96 to 100]
Statistical Analysis 1: Comparison: Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1; The primary immunogenicity endpoint, the seroprotection rate after one dose of either vaccine candidate in the OPV-vaccinated groups (nOPV2 combined groups 1 and 2, and combined groups 3 and 4), was compared with the corresponding endpoint from the historical monovalent OPV2 (mOPV2) control study (UAM1, EudraCT # 2015-003325-33). In the UAM1 study, the observed seroprotection rate after a single dose of mOPV2 was 98% (98 out of 100 participants), with a 95% confidence interval (CI) of 93-100%; Test type: Non-Inferiority — The primary immunogenicity endpoint, seroprotection on Day 28 after a single dose of each vaccine candidate, was formally compared with the corresponding endpoint from UAM1 via a non-inferiority test of the difference of each of the novel candidates to the monovalent OPV2 control, mOPV2, each using one-sided α=0.025 and a non-inferiority margin of 10%, computed using two-sided α=0·05 Miettinen and Nurminen score-based CIs for inference; Difference = 2.0, 95% CI 2-sided [-1.9 to 7.0]
Statistical Analysis 2: Comparison: Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2; The primary immunogenicity endpoint, the seroprotection rate after one dose of either vaccine candidate in the OPV-vaccinated groups (nOPV2 combined groups 1 and 2, and combined groups 3 and 4), was compared with the corresponding endpoint from the historical monovalent OPV2 control study (UAM1, EudraCT # 2015-003325-33). In the UAM1 study, the observed seroprotection rate after a single dose of mOPV2 was 98% (98 out of 100 participants), with a 95% confidence interval (CI) of 93-100%; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference = 2.0, 95% CI 2-sided [-1.8 to 7.0]

3. Secondary Outcome: Number of Former OPV Recipients With Solicited Adverse Events Within 7 Days of Vaccination With Novel OPV2
Description: Participants were asked to complete 7-day diary cards soliciting systemic adverse events and daily oral temperature. Solicited events comprised selected signs and symptoms including headache, fatigue, myalgia, arthralgia, paresthesia, anesthesia, paralysis, nausea, vomiting, diarrhea and abdominal pain, or fever defined as a temperature of 37.5°C or higher.
  AEs were graded as mild (easily tolerated with minimal discomfort or temperature 37.5°C to 38.0°C), moderate (sufficiently discomforting to interfere with normal everyday activities, or temperature 38.1°C to 39.0°C), or severe (preventing normal everyday activities, or temperatures higher than 39.0°C).
  AEs were assessed by the investigator for causality. Probably related suggests that a reasonable temporal sequence of the AE with vaccine administration exists and, in the Investigator's clinical judgment, it is likely that a causal relationship exists between the vaccine administration and the AE,
Time Frame: Up to 7 days after each dose (Day 0-7 post-dose 1 and Day 28-35 post-dose 2)
Population: Participants in the total vaccinated population previously vaccinated with OPV.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 1: Participants previously vaccinated with OPV received vaccination with novel OPV2 candidate 1 on study Day 0.
- Group 2: OPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 2: Participants previously vaccinated with OPV received a second vaccination with novel OPV2 candidate 1 on Day 28.
- Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 1: Participants previously vaccinated with OPV received vaccination with novel OPV2 candidate 2 on study Day 0.
- Group 4: OPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 2: Participants previously vaccinated with OPV received a second vaccination with novel OPV2 candidate 2 on Day 28.
Arm/Group | Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 1 | Group 2: OPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 2 | Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 1 | Group 4: OPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 2
Number analyzed (Participants) | 100 | 49 | 100 | 49
Participants
  Any solicited adverse event | 71 | 26 | 74 | 21
  Mild | 45 | 18 | 60 | 14
  Moderate | 23 | 8 | 12 | 6
  Severe | 3 | 0 | 2 | 1
  Probably related to vaccination | 44 | 15 | 37 | 12

4. Secondary Outcome: Number of Former IPV Recipients With Solicited Adverse Events After Vaccination With Novel OPV2
Description: as for outcome 3
Time Frame: 7 days post-dose (Day 0-7 post-dose 1 and and Day 28-35 post-dose 2)
Population: Participants in the total vaccinated population previously vaccinated with IPV only.
Measure: Count of Participants; unit: Participants
Groups:
- Group 5: IPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 1: Participants previously vaccinated with only IPV received a vaccination with novel OPV2 candidate 1 on Day 0.
- Group 5: IPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 2: Participants previously vaccinated with only IPV received a second vaccination with novel OPV2 candidate 1 on Day 28.
- Group 6: IPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 1: Participants previously vaccinated with only IPV received a vaccination with novel OPV2 candidate 2 on Day 0.
- Group 6: IPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 2: Participants previously vaccinated with only IPV received a second vaccination with novel OPV2 candidate 2 on Day 28.
- Group 7: IPV-vaccinated - Placebo Post-dose 1: Participants previously vaccinated with only IPV received a vaccination with placebo on Day 0.
- Group 7: IPV-vaccinated - Placebo Post-dose 2: Participants previously vaccinated with only IPV received a second vaccination with placebo on Day 28.
Arm/Group | Group 5: IPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 1 | Group 5: IPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 2 | Group 6: IPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 1 | Group 6: IPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 2 | Group 7: IPV-vaccinated - Placebo Post-dose 1 | Group 7: IPV-vaccinated - Placebo Post-dose 2
Number analyzed (Participants) | 17 | 17 | 16 | 15 | 17 | 16
Participants
  Any solicited adverse events | 16 | 11 | 13 | 9 | 15 | 12
  Mild | 11 | 8 | 6 | 3 | 9 | 7
  Moderate | 4 | 3 | 7 | 5 | 4 | 5
  Severe | 1 | 0 | 0 | 1 | 2 | 0
  Probably related to vaccination | 9 | 8 | 5 | 8 | 9 | 5

5. Secondary Outcome: Number of Participants With Unsolicited Adverse Events
Description: Unsolicited events comprised other signs and symptoms that participants reported through the end of the study. Each unsolicited AE was rated on a 3-point scale of increasing intensity:
  * Grade 1: Mild; an AE that was easily tolerated by the subject, causing minimal discomfort and not interfering with everyday activities.
  * Grade 2: Moderate; an AE that was sufficiently discomforting to interfere with normal everyday activities.
  * Grade 3: Severe; an AE that prevented normal everyday activities. Each adverse event was assessed by the investigator for causality as unrelated, unlikely, possibly, or probably related to the vaccination.
Time Frame: Up to 42 days after each vaccination
Population: Total vaccinated population
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Number analyzed (Participants) | 50 | 50 | 50 | 50 | 17 | 16 | 17
Participants
  Any unsolicited adverse event | 34 | 43 | 38 | 42 | 15 | 13 | 17
  Mild | 8 | 10 | 10 | 11 | 3 | 0 | 1
  Moderate | 18 | 18 | 24 | 24 | 8 | 8 | 7
  Severe | 8 | 15 | 4 | 7 | 4 | 5 | 9
  Probably related to vaccination | 2 | 2 | 1 | 2 | 1 | 2 | 1

6. Secondary Outcome: Number of Former OPV Recipients With Clinically Relevant Laboratory Abnormalities Up to 28 Days After Each Vaccination
Description: Laboratory assessments were collected at one-week intervals from Day 0 to Day 28 (except for Day 21) and at Days 35, 42, and 56 for participants in Groups 2 and 4 who received a 2nd dose.
  The Investigator reviewed laboratory values outside the normal range and assessed their clinical relevance.
  Any clinically relevant abnormal lab values that occurred at any visit up to 28 days after the first vaccination (in combined Groups 1 and 2 and Groups 3 and 4) and up to 28 days (Day 56) after the second dose (Groups 2 and 4) are reported.
Time Frame: Day 0, Day 7, Day 14, and Day 28 for Groups 1-4 and at Day 35, Day 42, and Day 56 for participants in Groups 2 and 4
Population: Participants in the total vaccinated population previously vaccinated with OPV.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 Post-dose 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2 Post-dose 1 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2
Number analyzed (Participants) | 100 | 50 | 100 | 50
Participants | 28 | 18 | 30 | 15

7. Secondary Outcome: Number of Former IPV Recipients With Clinically Relevant Laboratory Abnormalities Up to 28 Days After Each Vaccination
Description: Laboratory assessments were collected at one-week intervals from Day 0 to Day 56, except for Days 21 and 49. The Investigator reviewed laboratory values outside the normal range and assessed their clinical relevance.
  Any clinically relevant abnormal laboratory abnormalities that occurred at any visit up to 56 days are reported.
Time Frame: Day 0, Day 7, Day 14, Day 28, Day 35, Day 42 and Day 56
Population: Participants in the total vaccinated population previously vaccinated with IPV only.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Number analyzed (Participants) | 17 | 16 | 17
Participants | 4 | 6 | 9

8. Secondary Outcome: Anti-Poliovirus Type-2 Neutralizing Antibody Titers After A Single Dose of Novel OPV2
Description: Neutralizing antibodies against poliovirus type 2 were determined using the World Health Organization (WHO) standard microneutralization assay (WHO EPI GEN 93.9). The lower limit of quantitation (LLOQ) was 5.7 and the upper limit of quantitation (ULOQ) was 1448. Data were calculated on log2-transformed type 2 neutralizing titers and back transformed for the presentation below. Values shown as 1448 should be interpreted as ≥ 1448.
Time Frame: Day 0 and Day 28
Population: Per-protocol population. The per-protocol population excluded participants with missed doses or major protocol deviations considered to have a potential impact on immunogenicity from the time of the deviation and at all time points thereafter. This endpoint was analyzed after one dose of nOPV hence Groups 1 and 2 and Groups 3 and 4 are combined for analysis, as specified in the study protocol. Samples for 2 participants in Group 5 on Day 0 were mixed up and are not included in the analysis.
Measure: Median (Inter-Quartile Range); unit: titer
Groups:
- Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1: Participants previously vaccinated with OPV received a vaccination with novel OPV2 candidate 1 on study Day 0.
- Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2: Participants previously vaccinated with OPV received a vaccination with novel OPV2 candidate 2 on study Day 0.
- Group 5: IPV-vaccinated - Novel OPV2 Candidate 1: Participants previously vaccinated with only IPV received a vaccination with novel OPV2 candidate 1 on Day 0.
- Group 6: IPV-vaccinated - Novel OPV2 Candidate 2: Participants previously vaccinated with only IPV received a vaccination with novel OPV2 candidate 2 on Day 0.
- Group 7: IPV-vaccinated - Placebo: Participants previously vaccinated with only IPV received a vaccination with placebo on Day 0.
Arm/Group | Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 | Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Placebo
Number analyzed (Participants) | 98 | 98 | 17 | 16 | 16
titer
  Day 0 (pre-vaccination): number analyzed (Participants) | 98 | 98 | 15 | 16 | 16
  Day 0 (pre-vaccination) | 324 [228 to 455] | 455 [256 to 724] | 228 [74 to 588] | 144 [26 to 446] | 91 [11 to 362]
  Day 28: number analyzed (Participants) | 96 | 98 | 17 | 16 | 16
  Day 28 | 1448 [1448 to 1448] | 1152 [815 to 1448] | 1448 [1448 to 1448] | 1448 [1176 to 1448] | 51 [8 to 256]

9. Secondary Outcome: Seroprotection Rate 28 Days After Two Doses of Novel OPV2 in Former OPV Recipients
Description: Seroprotection rate was defined as the percentage of participants with anti-type 2-specific poliovirus neutralizing antibodies titers ≥ 1:8.
Time Frame: Day 56
Population: Participants in the per-protocol population previously vaccinated with OPV who received 2 doses of novel OPV2 (Groups 2 and 4).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2
Number analyzed (Participants) | 49 | 49
percentage of participants | 100 [93 to 100] | 100 [93 to 100]

10. Secondary Outcome: Seroprotection Rate in Former IPV Recipients
Description: as for outcome 9
Time Frame: Day 0, Day 28, and Day 56
Population: Participants in the per-protocol population previously vaccinated with IPV only. Samples for 2 participants in Group 5 on Day 0 were mixed up and are not included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Number analyzed (Participants) | 17 | 16 | 16
percentage of participants
  Day 0 (pre-vaccination): number analyzed (Participants) | 15 | 16 | 16
  Day 0 (pre-vaccination) | 93 [68 to 100] | 94 [70 to 100] | 81 [54 to 96]
  Day 28 | 100 [80 to 100] | 100 [79 to 100] | 75 [48 to 93]
  Day 56: number analyzed (Participants) | 17 | 15 | 16
  Day 56 | 100 [80 to 100] | 100 [78 to 100] | 81 [54 to 96]

11. Secondary Outcome: Seroconversion Rate After a Single Dose of Novel OPV2 in Former OPV Recipients
Description: Seroconversion is defined as a change from seronegative to seropositive (poliovirus type-2-specific neutralizing antibody titers ≥ 1:8), or for participants seropositive at Baseline, an antibody titer increase of ≥ 4-fold over Baseline titer.
Time Frame: Day 28
Population: Participants in the seroconversion subset of the per-protocol population previously vaccinated with OPV. The seroconversion subset included participants with Baseline titer sufficiently low to enable observation of a four-fold increase without breaching the ULOQ (ie, a titer ≤ 362).
  Since this endpoint was analyzed after 1 dose of nOPV, Groups 1 and 2 and Groups 3 and 4 are combined for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1+2: OPV-vaccinated - Novel OPV2 Candidate 1 | Group 3+4: OPV-vaccinated - Novel OPV2 Candidate 2
Number analyzed (Participants) | 55 | 47
percentage of participants | 74.5 [61.0 to 85.3] | 51.1 [36.1 to 65.9]

12. Secondary Outcome: Seroconversion Rate After Two Doses of Novel OPV2 in Former OPV Recipients
Description: as for outcome 11
Time Frame: Day 56
Population: Participants in the seroconversion subset of the per-protocol population previously vaccinated with OPV and who received 2 doses of novel OPV2 (Groups 2 and 4). The seroconversion subset included participants with Baseline titer sufficiently low to enable observation of a four-fold increase without breaching the ULOQ (ie, a titer ≤ 362).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2
Number analyzed (Participants) | 27 | 26
percentage of participants | 74 [54 to 89] | 58 [37 to 77]

13. Secondary Outcome: Seroconversion Rate in Former IPV Recipients
Description: Seroconversion is defined as a change from seronegative to seropositive (poliovirus type-2-specific neutralizing antibody titers ≥ 1:8), or for participants seropositive at Baseline, a poliovirus type-2-specific neutralizing antibody titer increase of ≥ 4-fold over Baseline titer.
Time Frame: Day 28 and Day 56
Population: Participants in the seroconversion subset of the per-protocol population previously vaccinated with IPV only. The seroconversion subset included participants with Baseline titer sufficiently low to enable observation of a four-fold increase without breaching the ULOQ (ie, a titer ≤ 362).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
Number analyzed (Participants) | 10 | 12 | 12
percentage of participants
  Day 28 | 100 [69 to 100] | 92 [62 to 100] | 0 [0 to 26]
  Day 56: number analyzed (Participants) | 10 | 11 | 12
  Day 56 | 100 [69 to 100] | 82 [48 to 98] | 8 [0 to 38]

ADVERSE EVENTS:
Time Frame: Up to 42 days after each vaccination (42 days in Groups 1 and 3 and 70 days for all other Groups).
Groups:
- Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2: Participants previously vaccinated OPV received two doses of novel OPV2 candidate 2 28 days apart (Day 0 and Day 28).
Arm/Group | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 | Group 7: IPV-vaccinated - Two Doses of Placebo
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50 | 0/50 | 0/50 | 0/17 | 0/16 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/50 | 1/50 | 0/50 | 1/50 | 0/17 | 1/16 | 0/17
Other Adverse Events (participants affected / at risk) | 44/50 | 48/50 | 47/50 | 47/50 | 17/17 | 15/16 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 (N=50) | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 (N=50) | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 (N=50) | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 (N=50) | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 (N=17) | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 (N=16) | Group 7: IPV-vaccinated - Two Doses of Placebo (N=17)
Crohn's Disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: OPV-vaccinated - One Dose of Novel OPV2 Candidate 1 (N=50) | Group 2: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 (N=50) | Group 3: OPV-vaccinated - One Dose of Novel OPV2 Candidate 2 (N=50) | Group 4: OPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 (N=50) | Group 5: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 1 (N=17) | Group 6: IPV-vaccinated - Two Doses of Novel OPV2 Candidate 2 (N=16) | Group 7: IPV-vaccinated - Two Doses of Placebo (N=17)
Upper Respiratory Tract Infection (Infections and infestations) | 9 | 4 | 7 | 13 | 0 | 5 | 9
Nasopharyngitis (Infections and infestations) | 4 | 4 | 1 | 2 | 5 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 1 | 1 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 3 | 0 | 0 | 1 | 2 | 0
Oral Herpes (Infections and infestations) | 0 | 2 | 0 | 1 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 1 | 1 | 1 | 2 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acute Sinusitis (Infections and infestations) | 1 | 1 | 0 | 1 | 2 | 0 | 0
Enterobiasis (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis Viral (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Oral Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tinea Pedis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viral Rhinitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 11 | 14 | 16 | 14 | 6 | 5 | 7
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 2 | 0 | 4 | 2
Migraine (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Sleep Deficit (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 4 | 3 | 3 | 6 | 6 | 3 | 3
Abdominal Pain (Gastrointestinal disorders) | 0 | 3 | 3 | 4 | 1 | 2 | 4
Nausea (Gastrointestinal disorders) | 0 | 3 | 5 | 1 | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 0 | 0 | 0
Aphthous Ulcer (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 3 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 3 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Gastrointestinal Sounds Abnormal (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dental Caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia Teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rectal Tenesmus (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Swollen Tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tongue Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 8 | 7 | 5 | 3 | 1 | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 3 | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 3 | 2 | 0 | 0 | 3 | 3
Influenza Like Illness (General disorders) | 1 | 3 | 4 | 1 | 1 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Malaise (General disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 1
Hangover (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Chest Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Crepitations (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Feeling Cold (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Feeling Hot (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3 | 1 | 0 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 2 | 0 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 3 | 0 | 1 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 3 | 1 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 3 | 5 | 4 | 5 | 1 | 0 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 1 | 0 | 1 | 0 | 0 | 1
C-Reactive Protein Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 1
Neutrophil Count Increased (Investigations) | 0 | 1 | 1 | 1 | 0 | 0 | 0
Blood Immunoglobulin A Decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Blood Potassium Increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Lymphocyte Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte Percentage Decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 4 | 3 | 5 | 0 | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 1
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Rash Generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 3 | 0 | 1 | 2 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 3 | 1 | 0 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Animal Bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Procedural Nausea (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Procedural Pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Middle Ear Disorder (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Burnout Syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Irritation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear Lobe Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Herpes Zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash Pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tension Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abnormal Faeces (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eosinophil Count Increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Platelet Count Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04544787/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT04544787/SAP_001.pdf